CLINICAL TRIAL: NCT00005770
Title: Investigation of the Effect of Acupuncture Needling on Connective Tissue Using Ultrasound Elastography
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Other Study IDs: NCRR-M01RR00109-0745; M01RR000109 (NIH)
Record Dates: First submitted 2000-06-01; First posted 2000-06-02 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-11

CONDITIONS: Healthy
Keywords: elastic property of skin
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Cross-Sectional

INTERVENTIONS:
Device: Acupuncture

SUMMARY:
During acupuncture treatment, acupuncture needles are inserted and manipulated until a characteristic local tissue reaction termed "de qi" is observed. De qi can be perceived by the acupuncturist in the form of "needle grasp", a mechanical gripping of the needle by the tissue. De qi is considered essential to the therapeutic effect of acupuncture. Therefore, the investigator proposes that understanding this local tissue reaction will lead to an understanding of how the therapeutic effect of acupuncture therapy arises. Specifically, it is hypothesized that needle manipulation causes winding of collagen and elastic fibers around the needle. This action induces tension in the collagen network surrounding the needling site and results in a mechanical signal that is transduced into local cells. The objective of the current work is to use ultrasound elastography, a recently developed ultrasound imaging technique, to visualize and quantify changes in the elastic properties of skin and subcutaneous tissue in 12 healthy human volunteers as a result of acupuncture needle manipulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont, Burlington, Vermont, United States